CLINICAL TRIAL: NCT00447135
Title: Immunologic Function in the Elderly After Injury: the Polymorphonuclear Leukocyte (PMN) and Innate Immunity
Brief Title: Immunologic Function in the Elderly After Injury
Status: Completed | Type: Observational
Sponsor: Summa Health System (Other)
Responsible Party: Dr. William Fallon, Summa Health System
Other Study IDs: 04104
Record Dates: First submitted 2006-08-07; First posted 2007-03-14 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2008-01

CONDITIONS: Over the Age of 65; Admitted to the Trauma Service
Keywords: Elderly; Trauma; Polymorphonuclear Leukocyte; Immunity
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research is to learn more about the function of the body's ability to fight infection when the immune response is activated when injury occurs, in the elderly population.

DETAILED DESCRIPTION:
Injury in the elderly is characterized by higher mortality rates, longer hospital stays and increased long term disability when controlled for injury severity as compared to the younger cohort of injury patients.(7) The greater likelihood of co-morbid, pre-existing medical conditions, which have a negative impact on outcome, may in part be responsible for this observation. However, there is some disagreement about whether there is an impact of physiologic age as opposed to chronological age on outcomes and whether this is the most important determining factor for the injured elderly. (8) It is clear that the combination of an age factor and baseline health status may determine the ability of the elderly injured patient to recover successfully. This may be due to age related degradation in immune function either PMN related or cell mediated immunity (CMI) related.

In healthy individuals, the metabolic response to hemorrhage, burns and injury is characterized by a hyperdynamic metabolic response that upregulates the proinflammatory/immunologic/metabolic "milieu" and is designed to heal injury, combat infection and prevent death. This inflammatory response on the part of the patient is both functional and adaptive from a physiologic perspective (9). Aging is known to decrease physiologic reserve and may play a role in altering the ability of the injured elderly patient to mount an adaptive, appropriate, inflammatory response when injured (10). Some evidence exists that documents the age-related decline of immunologic function in the elderly, particularly that portion of the immune response described as cell mediated immunity [CMI] (11). This contributes to the higher increase in infections in the elderly (12). There is also animal model evidence that immune function is worsened when combined with injury (13). Similarly, hemorrhage, burns and injury also depress cell mediated immunity in previously healthy individuals increasing the likelihood of infection and organ system failure as a result (14). Little is known, however, about the nature of the immuno/inflammatory response to injury in the elderly. Therefore, one of the hypotheses of our study is that the aging process attenuates this immuno/inflammatory response process, adversely impacting the function of the nonspecific portion of the immune defense system and the main component of that system, the polymorphonuclear leukocyte (PMN).

The systemic immuno/inflammatory response to hemorrhage, burns and injury is well characterized in young, healthy volunteers and animal models and has been studied extensively (15). The key feature of this response is the attraction of PMNs to the site of injury. These are "mature" PMNs that are present in the peripheral bloodstream that possess a life span of approximately 3-5 days. When activated, these cells are responsible for limiting microbial invasion and promoting wound healing. However, prolonged activation of these cells is deleterious as it can lead to perpetuation of the inflammatory response, exacerbating tissue injury and leading to the development of organ system injury, and the condition known as multi-system organ failure. Under normal circumstances, the process of apoptosis, or programmed cellular death, limits the life span of the PMN to 2-3 days and serves to regulate the extent of the immuno/inflammatory response. This allows sufficient time for the acquired immune system to be activated and come on line in response to the cell mediated activity against infection and antigen. Many of the normal functions of the innate, non-specific PMN dependent, immune system are known to be dysfunctional in younger patients who have sepsis, severe injury or shock. It is unclear, however, if the same impact is present in elderly patients who have been injured because little is known about the function of the PMNs in elderly patients in general, and, specifically in those elderly patients who have been injured. Since elderly patients have known, age related depressed cell mediated immunity, our second hypothesis is that there may be age related abnormalities present in the PMNs of elderly patients who have been injured that contribute to the worse outcomes following injury.

The purpose of this study is to begin to characterize the functional status of a portion of the innate immune response following injury in elderly trauma patients. This will be accomplished through analysis of a standard battery of functional tests that characterize PMNs regarding apoptosis and responses to immune challenges. These PMN functionality tests will be correlated with observed clinical outcomes. The null hypothesis for this study is that PMNs from elderly trauma patients have functional characteristics that result in different local and systemic effects than PMN's from non-injured elder controls or non-injured non-elder controls and that this may lead to different effects post injury that impact outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 65
* Admitted to the trauma service

Exclusion Criteria:

* Inability to draw sufficient blood
* Immunocompromised
* Currently receiving systemic corticosteroids
* Participation in other studies
* In the opinion of the investigator will not be able to complete protocol

Min Age: 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Elderly after injury
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2005-03; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Fallon, MD, Principal Investigator — Summa Health System
Locations (1):
- Summa Health System, Akron, Ohio, United States